CLINICAL TRIAL: NCT03877822
Title: The Impact of Two Days of Bed Rest Versus Two Days of Habitual Activity on Insulin Sensitivity and Cumulative Muscle Protein Synthesis in Healthy Young Males
Brief Title: Two-day Bed Rest, Insulin Sensitivity and Muscle Protein Synthesis
Acronym: 2d-BR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study protocol no longer relevant after progression of the scientific field
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 190206/B/05
Record Dates: First submitted 2019-02-28; First posted 2019-03-18 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Healthy
MeSH Terms: interventions — Bed Rest

STUDY DESIGN:
Intervention Model Description: Participants will firstly undergo 2 days of habitual physical activity, followed by 2 days of bed rest
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Habitual activity and 2 days bed rest (Experimental): Participants will undergo 2 days of habitual activity and 2 days bed rest
  Interventions: Behavioral: Habitual activity; Behavioral: Bed rest

INTERVENTIONS:
Behavioral: Habitual activity — Two days of habitual physical activity, under normal free-living conditions
Behavioral: Bed rest — Two days of bed rest, to induce whole-body physical inactivity

SUMMARY:
The impact of two days bed rest versus two days of habitual activity on insulin sensitivity and cumulative muscle protein synthesis will be investigated in healthy young males

DETAILED DESCRIPTION:
To study the mechanisms underlying inactivity-induced muscle atrophy, the impact of two days bed rest versus two days of habitual activity on insulin sensitivity and cumulative muscle protein synthesis will be investigated in healthy young males

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18-40

Exclusion Criteria:

* Smoker
* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes)
* Any diagnosed cardiovascular disease (e.g. deep vein thrombosis or hypertension)
* Chronic use of any prescribed or over the counter pharmaceuticals (that may modulate muscle protein metabolism).
* A personal or family history of thrombosis, epilepsy, seizures or schizophrenia.
* Any known disorders in muscle metabolism
* Regular use of nutritional supplements (i.e. ingestion more than twice per week during the last month)
* Metallic implants (including heart pacemaker, cochlear implants, medication pumps, surgical clips, plates or screws).
* Allergy to lidocaine
* Recent (within the last 6 months) or current musculoskeletal injury (e.g. leg fracture)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in whole-body insulin sensitivity | During 2 days of habitual physical activity and 2 days of bed rest. Blood glucose and insulin are monitored for 2 hours following ingestion of a standardized meal
  Change in whole-body insulin sensitivity via meal tolerance test

SECONDARY OUTCOMES:
Change in cumulative muscle protein synthesis | During 2 days of habitual physical activity and 2 days of bed rest
  Cumulative muscle protein synthesis via deuterium oxide ingestion. The incorporation of deuterated alanine in muscle is expressed relative to body water enrichments, to obtain muscle protein synthesis in %/day
Change in continuous glucose | Continuous glucose, during the 2 days of habitual activity and 2 days of bed rest
  Change in continuous glucose via continuous glucose monitoring.
Change in muscle volume | Immediately before and immediately after the 2-day bed rest period
  Change in muscle volume via MRI

CONTACTS AND LOCATIONS:
Overall Officials: Marlou L Dirks, PhD, Principal Investigator — University of Exeter